CLINICAL TRIAL: NCT04428411
Title: The Impact of Difficult to Treat Sites on Biological Treatment Response in Patients With Moderate-to-Severe Plaque Psoriasis
Brief Title: Study To Evaluate The Impact Of Difficult To Treat Sites On Biological Response In Moderate-To-Severe Plaque Psoriasis(PsO).
Status: Completed | Type: Observational
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: B1801416
Record Dates: First submitted 2020-06-10; First posted 2020-06-11 (Actual); Results first posted 2021-10-25 (Actual); Last update posted 2021-10-25 (Actual); Status verified 2021-09

CONDITIONS: Plaque Psoriasis
MeSH Terms: interventions — Etanercept

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with moderate to severe plaque psoriasis: Iraqi patients diagnosed with moderate to severe plaque psoriasis that received Enbrel as treatment for disease
  Interventions: Drug: Enbrel

INTERVENTIONS:
Drug: Enbrel — As provided in real world practice

SUMMARY:
This study is to evaluate available local data in Iraq patients with moderate-to-severe plaque psoriasis on Enbrel treatment with regards to efficacy, treatment for PsO who have difficult to treat sites at presentation.

ELIGIBILITY:
Inclusion Criteria:

* Moderate-to-severe plaque psoriasis patients whom have been receiving etanercept for at least 1 year duration.
* Have difficult to treat sites at presentation.
* Age ≥18 years.
* No history of using other biological treatments, other than etanercept for the treatment of moderate-to-severe PsO.

Exclusion Criteria:

* Etanercept use for treatment of moderate-to-severe PsO less than 1 year duration.
* Previous use of another biological treatment for treatment of moderate-to-severe PsO.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients data from the local Dermatology Center of the Baghdad Teaching Hospital
Sampling Method: Non-Probability Sample
Enrollment: 486 (Actual)
Dates: Start 2020-07-05 (Actual); Primary Completion 2020-08-30 (Actual); Study Completion 2020-08-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (1):
- Pfizer, Baghdad, Iraq

IPD SHARING:
Plan to Share IPD: No
Pfizer will provide access to individual de-identified participant data and related study documents (e.g. protocol, Statistical Analysis Plan (SAP), Clinical Study Report (CSR)) upon request from qualified researchers, and subject to certain criteria, conditions, and exceptions. Further details on Pfizer's data sharing criteria and process for requesting access can be found at: https://www.pfizer.com/science/clinical_trials/trial_data_and_results/data_requests.

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://pmiform.com/clinical-trial-info-request?StudyID=B1801416

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Data of Iraq's participants aged greater than or equal to (>=) 18 years, who received etanercept for at least 1 year (from August 2015 to April 2020) for treatment of moderate to severe psoriasis were included in the study. Data source was the local registry at dermatology center of Baghdad teaching hospital. Available data were evaluated for approximately 1.8 months for this retrospective, observational study.
Groups:
- Etanercept: Participants received etanercept to treat moderate-to severe plaque psoriasis for at least 1 year from August 2015 to April 2020 under real world standard clinical practice (in Iraq, the recommended dose of etanercept [Enbrel] is 25 milligrams [mg] administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied in this observational study.
Period: Overall Study
Arm/Group | Etanercept
Started | 486
Participants With Difficult to Treat Sites | 397
Participants Without Difficulty to Treat Sites | 89
Participants Adherent to Treatment | 417
Participants Not Adherent to Treatment | 69
Completed | 372
Not Completed | 114
Not completed — Lost to Follow-up | 114

BASELINE CHARACTERISTICS:
Population: Analysis was performed on all participants whose data were included in the study for retrospective observation.
Groups:
- Etanercept: Participants received etanercept to treat moderate-to severe plaque psoriasis for at least 1 year from August 2015 to April 2020 under real world standard clinical practice (in Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly). Data of these participants were studied in this observational study.
Arm/Group | Etanercept
Number analyzed (Participants) | 486
Age, Continuous [Mean (Standard Deviation); unit: Years] | 32.5 (10.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 246
  Male | 240
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Disease duration [Mean (Standard Deviation); unit: Years] | 10.6 (6.4)

OUTCOME MEASURES:

1. Primary Outcome: Mean Change From Baseline in Percent Body Surface Area (BSA) Score at Month 4
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area of a body region was counted. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint equal to (=) 10 percent (%) for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%. Higher % BSA = greater severity of psoriasis. This outcome measure evaluated comparison between participants with and without difficulty to treat sites.
Time Frame: Baseline (pre-treatment), Month 4 (post-treatment) (from the data retrieved and observed in approximately 1.8 months of this study)
Population: Analysis was performed on all participants whose data were included in the study for retrospective observation. Here, "Number Analyzed" signifies participants evaluable at specific time points.
Measure: Mean (Standard Deviation); unit: Percent BSA
Groups:
- Etanercept: Participants With Difficult to Treat Sites: Participants received etanercept to treat moderate-to severe plaque psoriasis for at least 1 year from August 2015 to April 2020 under real world standard clinical practice (in Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly) and had sites difficult to treat.
- Etanercept: Participants Without Difficult to Treat Sites: Participants received etanercept to treat moderate-to severe plaque psoriasis for at least 1 year from August 2015 to April 2020 under real world standard clinical practice (in Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly) and did not have sites difficult to treat.
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 397 | 89
Percent BSA
  Baseline | 28.1 (19.603) | 29.21 (18.757)
  Change at Month 4: number analyzed (Participants) | 391 | 89
  Change at Month 4 | -6.79 (17.472) | -6.38 (17.012)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p = 0.35, t-test, 2 sided

2. Primary Outcome: Mean Change From Baseline in Percent Body Surface Area (BSA) Score at Month 12
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area of a body region was counted. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint = 10 % for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%. Higher % BSA = greater severity of psoriasis. This outcome measure evaluated comparison between participants with and without difficulty to treat sites.
Time Frame: Baseline (pre-treatment), Month 12 (post-treatment) (from the data retrieved and observed in approximately 1.8 months of this study)
Population: Analysis was performed on all participants whose data were included in the study for retrospective observation. Here, "Overall Number of Participants Analyzed" signifies participants evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: Percent BSA
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 344 | 78
Percent BSA | -19.13 (17.451) | -18.93 (16.555)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p = 0.07, t-test, 2 sided

3. Primary Outcome: Mean Change From Baseline in Percent Body Surface Area (BSA) Score at Last Visit
Description: as for outcome 2
Time Frame: Baseline (pre-treatment), Last Visit (any time after 12 months till maximum of approximately 5 years) (from the data retrieved and observed in approximately 1.8 months of this study)
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent BSA
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 300 | 72
Percent BSA | -23.78 (17.799) | -24.4 (16.876)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p = 0.41, t-test, 2 sided

4. Primary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Month 4
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants. This outcome measure evaluated comparison between participants with and without difficulty to treat sites.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 397 | 89
Units on a scale
  Baseline | 24.6 (4.303) | 24.42 (4.014)
  Change at Month 4: number analyzed (Participants) | 391 | 89
  Change at Month 4 | -5.75 (5.306) | -7.56 (5.797)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p = 0.01, t-test, 2 sided

5. Primary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Month 12
Description: as for outcome 4
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 344 | 78
Units on a scale | -15.66 (6.299) | -17.39 (5.442)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p = 0.02, t-test, 2 sided

6. Primary Outcome: Mean Change From Baseline in Dermatology Life Quality Index (DLQI) Score at Last Visit
Description: as for outcome 4
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 300 | 72
Units on a scale | -17.49 (6.204) | -19.39 (4.604)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p = 0.09, t-test, 2 sided

7. Primary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Month 4
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 (no disease) to 72.0 (maximum disease), with higher scores representing greater severity of psoriasis. This outcome measure evaluated comparison between participants with and without difficulty to treat sites.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 397 | 89
Units on a scale
  Baseline | 24.68 (9.023) | 21.46 (10.621)
  Change at Month 4: number analyzed (Participants) | 391 | 89
  Change at Month 4 | -8.22 (9.224) | -6.22 (10.572)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p = 0.31, t-test, 2 sided

8. Primary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Month 12
Description: as for outcome 7
Time Frame: as for outcome 2
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on a scale
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 344 | 78
Units on a scale | -17.68 (7.934) | -16.16 (9.334)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p < 0.05, t-test, 2 sided

9. Primary Outcome: Mean Change From Baseline in Psoriasis Area and Severity Index (PASI) Score at Last Visit
Description: as for outcome 7
Time Frame: as for outcome 3
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept: Participants With Difficult to Treat Sites | Etanercept: Participants Without Difficult to Treat Sites
Number analyzed (Participants) | 300 | 72
Units on scale | -19.79 (7.922) | -18.42 (9.472)
Statistical Analysis 1: Comparison: Etanercept: Participants With Difficult to Treat Sites vs Etanercept: Participants Without Difficult to Treat Sites; Test type: Other; p < 0.05, t-test, 2 sided

10. Secondary Outcome: Percent Body Surface Area (BSA) Score at Baseline, Month 4, and Month 12 in Participants Adherent and Not Adherent to Treatment
Description: Four body regions were evaluated: head and neck, upper limbs, trunk (including axillae and groin) and lower limbs (including buttocks). Scalp, palms and soles were excluded. BSA was calculated using handprint method. Number of handprints (size of participant's full palmer hand) fitting in affected area of a body region was counted. Maximum number of handprints were 10 for head and neck, 20 for upper limbs, 30 for trunk and 40 for lower limbs. Surface area of body region equivalent to 1 handprint: 1 handprint = 10 percent (%) for head and neck, 5% for upper limbs, 3.33% for trunk and 2.5% for lower limbs. Percent BSA for a body region = total number of handprints in a body region * % surface area equivalent to 1 handprint. Overall % BSA for an individual: arithmetic mean of % BSA of all 4 body regions, ranged from 0 to 100%. Higher % BSA = greater severity of psoriasis. This outcome measure evaluated comparison between participants adherent and not adherent to treatment.
Time Frame: Baseline (pre-treatment), Month 4, 12 (post-treatment) (from the data retrieved and observed in approximately 1.8 months of this study)
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Percent BSA
Groups:
- Etanercept: Participants Adherent to Treatment: Participants received etanercept to treat moderate-to severe plaque psoriasis for at least 1 year from August 2015 to April 2020 under real world standard clinical practice (in Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly) and were adherent to treatment.
- Etanercept: Participants Not Adherent to Treatment: Participants received etanercept to treat moderate-to severe plaque psoriasis for at least 1 year from August 2015 to April 2020 under real world standard clinical practice (in Iraq, the recommended dose of etanercept [Enbrel] is 25 mg administered twice weekly or 50 mg administered once weekly. Alternatively, 50 mg given twice weekly might be used for up to 12 weeks followed, if necessary, by a dose of 25 mg twice weekly or 50 mg once weekly) and were not adherent to treatment.
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 417 | 69
Percent BSA
  Baseline | 27.56 (19.030) | 32.84 (21.324)
  Month 4: number analyzed (Participants) | 417 | 63
  Month 4 | 20.06 (11.706) | 31.74 (21.892)
  Month 12: number analyzed (Participants) | 353 | 69
  Month 12 | 8.7 (6.8) | 11.1 (8.9)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Comparison between Baseline and Month 4; Test type: Other; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Comparison between Baseline and Month 12; Test type: Other; p = 0.0001, t-test, 2 sided

11. Secondary Outcome: Dermatology Life Quality Index (DLQI) Score at Baseline, Month 4 and Month 12 in Participants Adherent and Not Adherent to Treatment
Description: DLQI is a 10-item questionnaire that measures the impact of skin disease on participant's quality of life over the last week. Each question was evaluated on a 4-point scale ranging from 0 (not at all) to 3 (very much); where higher scores indicated more impact on quality of life. Scores from all 10 questions added up to give DLQI total score range from 0 (not at all) to 30 (very much). Higher scores indicated more impact on quality of life of participants. This outcome measure evaluated comparison between participants adherent and not adherent to treatment.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 417 | 69
Units on scale
  Baseline | 24.50 (4.438) | 24.94 (2.838)
  Month 4: number analyzed (Participants) | 417 | 63
  Month 4 | 16.63 (6.303) | 21.19 (6.886)
  Month 12: number analyzed (Participants) | 353 | 69
  Month 12 | 6.6 (4.5) | 11.3 (7.2)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Comparison between Baseline and Month 4; Test type: Other; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Comparison between Baseline and Month 12; Test type: Other; p = 0.0001, t-test, 2 sided

12. Secondary Outcome: Psoriasis Area and Severity Index (PASI) Score at Baseline, Month 4, and Month 12 in Participants Adherent and Not Adherent to Treatment
Description: The PASI quantifies the severity of a participant's psoriasis based on both, "lesion severity" and the "percent of BSA" affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks]), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 (no disease) to 72.0 (maximum disease), with higher scores representing greater severity of psoriasis. This outcome measure evaluated comparison between participants adherent and not adherent to treatment.
Time Frame: as for outcome 10
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Units on scale
Arm/Group | Etanercept: Participants Adherent to Treatment | Etanercept: Participants Not Adherent to Treatment
Number analyzed (Participants) | 417 | 69
Units on scale
  Baseline | 21.980 (10.0055) | 22.458 (12.6765)
  Month 4: number analyzed (Participants) | 417 | 63
  Month 4 | 14.520 (8.8686) | 21.717 (15.8263)
  Month 12: number analyzed (Participants) | 353 | 69
  Month 12 | 4.8 (3.9) | 9.7 (6.4)
Statistical Analysis 1: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Comparison between Baseline and Month 4; Test type: Other; p = 0.0001, t-test, 2 sided
Statistical Analysis 2: Comparison: Etanercept: Participants Adherent to Treatment vs Etanercept: Participants Not Adherent to Treatment; Comparison between Baseline and Month 12; Test type: Other; p = 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Not applicable as adverse events were not collected for the study
Description: Due to non-interventional nature of study, the minimum criteria for reporting an adverse event (i.e., identifiable participant, identifiable reporter, a suspect product, and event) could not meet, hence adverse events were not collected and reported.
Arm/Group | Etanercept
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-07-27): https://cdn.clinicaltrials.gov/large-docs/11/NCT04428411/Prot_SAP_000.pdf